CLINICAL TRIAL: NCT07032714
Title: MAGENTA: Phase I Study of Mezigdomide and Talquetamab in Relapsed and Refractory Multiple Myeloma
Brief Title: Mezigdomide and Talquetamab in Relapsed and Refractory Multiple Myeloma
Acronym: MAGENTA
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Celgene Corporation (Industry); Janssen Research and Development LLC (Unknown)
Responsible Party: Principal Investigator, Andrew Yee, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-320
Record Dates: First submitted 2025-06-16; First posted 2025-06-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Relapsed Refractory Multiple Myeloma (RRMM)
Keywords: Relapsed Refractory Multiple Myeloma (RRMM); Prior therapy; Triple class exposed RRMM
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Cycle 1: Talquetamab and dexamethasone at a pre-determined escalating dose of talquetamab.
  Talquetamab is subcutaneously injected on Day 1, 4, 8, and 15 of the 28-day cycle. Dexamethasone is administered orally before receiving talquetamab (Days 1, 4, 8, 15).
  Cycle 2+: Mezigdomide, talquetamab, and dexamethasone Talquetamab is administered on Day 1 and 15 of cycles 2-6 and on Day 1 of cycles 7-12.
  Mezigdomide is administered orally once per day on days 1-21 of each 28-day cycle starting with cycle 2. This can continue until disease progression or withdrawal.
  Dexamethasone is administered orally once per week starting on Day 1 of Cycle 2 through cycle 6; the weekly dose will be split into 2 days.
  Interventions: Drug: Talquetamab; Drug: Mezigdomide; Drug: Dexamethasone
- Cohort B (Experimental): Cohort B takes place after Cohort A. Pre-phase 7 day cycle: Mezigdomide is administered orally once per day on Days 1-7. Dexamethasone is administered orally on Days 1 and 2.
  Cycle 1 (28 day cycle): Talquetamab is subcutaneously injected on Day 1, 4, 8, and 15 at a pre-determined escalating dose. Mezigdomide is given orally on days 1-14. Dexamethasone is administered orally as pre-medications before receiving talquetamab.
  Cycle 2+ (28 day cycle): Talquetamab on Days 1 and 15 of cycles 2-6; then Day 1 of cycles 7-12. Mezigdomide on Days 1-21 of cycles 2+ until disease progression or withdrawal. Dexamethasone on Days 1, 2, 8, 9, 15, 16, 22, 23 of cycles 2-6.
  Interventions: Drug: Talquetamab; Drug: Mezigdomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Talquetamab — Talquetamab is injected under the skin (subcutaneously injected) by trained medical staff. During first cycle of talquetamab, the dose of talquetamab will increase until the goal dose (treatment dose) is reached (pre-determined dose escalation).
Drug: Mezigdomide — Administered orally once per day (days 1-21 of applicable 28-day cycles; Days 1-7 of the 7-day Cohort B pre-phase cycle).
Drug: Dexamethasone — Administered orally once per day, at the schedule outlined in the Arm Descriptions.

SUMMARY:
This is a phase 1 study to find the recommended dose and schedule of mezigdomide and talquetamab in relapsed and refractory multiple myeloma (RRMM), and to test the effects of the drugs on cancer. Cohort A will receive talquetamab + dexamethasone, then mezigdomide + talquetamab,+ dexamethasone. After Cohort A, Cohort B will evaluate mezigdomide + dexamethasone followed by step-up dosing of talquetamab (mezigdomide + talquetamab,+ dexamethasone).

DETAILED DESCRIPTION:
This phase 1 open-label study will determine the recommended dose and schedule of mezigdomide and talquetamab in triple class exposed relapsed and refractory multiple myeloma. This study aims to enroll 25 participants including Cohorts A and B, and will follow a dose escalation schedule. Treatment is until progression or withdrawal of consent. The U.S. Food and Drug Administration (FDA) has not approved the combination of drugs mezigdomide, talquetamab, and dexamethasone as treatment for any disease. The FDA has not approved mezigdomide as a treatment for any disease. The FDA has approved talquetamab for the treatment of relapsed refractory multiple myeloma in patients who have already received 4 prior lines of therapy. Dexamethasone is approved by the FDA to treat multiple diseases including multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Participant has given voluntary signed written informed consent before performance of any study-related procedure that is not part of normal medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to their future medical care.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (see Appendix).
* Age ≥ 18 years
* Measurable disease of multiple myeloma as defined by at least one of the following:

  * Serum monoclonal protein ≥ 0.5 g/dL. Patients with IgD disease and lower amounts of monoclonal protein may be permitted to enroll with PI approval
  * ≥ 200 mg of monoclonal protein in the urine on 24-hour urine protein electrophoresis
  * Serum free light chain (FLC) ≥ 100 mg/L (10 mg/dL) and abnormal serum free light chain ratio
* Previously treated relapsed and refractory multiple myeloma:

  * Patients must have received at least three prior lines of therapy;
  * Prior therapy including an immunomodulatory drug, proteasome inhibitor, and anti-CD38 antibody (either in separate regimens or within the same regimen); and
  * Disease progression on, or within 60 days of completion of last therapy.
* ANC ≥ 1000/μL. G-CSF is not permitted within 14 days of screening.
* Platelet count ≥ 50,000/µL. Platelet transfusion and thrombopoietin receptor agonists are not permitted within 7 days of screening.
* Hemoglobin ≥ 8 g/dL. Red blood cell transfusions are permitted to meet eligibility criteria.
* Calculated creatinine clearance of ≥ 30 mL/min by Modified Diet in Renal Disease (MDRD) formula or Cockcroft-Gault formula
* Serum bilirubin values < 1.5 x ULN. Isolated bilirubin x 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%. Patients with elevated bilirubin due to Gilbert's syndrome may be permitted with PI approval (e.g. total bilirubin <3 mg/dL and normal direct bilirubin); and
* Serum aspartate transaminase (ALT) and aspartate transaminase (AST) values < 2.5 × the upper limit of normal (ULN) of the institutional laboratory reference range.
* Must be able to comply with thromboembolism prophylaxis with e.g. acetylsalicylic acid (ASA), apixaban, rivaroxaban, lower molecular weight heparin, or equivalent.
* Females of childbearing potential (FCBP) must:

  * Have 2 negative pregnancy tests as verified by the Investigator prior to starting study therapy. The subject must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.
  * Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use and be able to comply with two reliable forms of contraception as defined by the Pregnancy Prevention Plan.
* Male subjects must follow the mezigdomide Pregnancy Prevention Plan (see Appendix).
* Agree to follow the lifestyle considerations in Section 3.4 regarding blood donation, hospitalization and being in proximity to the hospital, and driving or operating heavy machinery.

Exclusion Criteria:

* Participants who have had myeloma therapy or investigational drug within 2 weeks prior to start of treatment or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Participants who are receiving any investigational agents.
* Prior therapy with mezigdomide or iberdomide.
* Prior therapy with anti-GPRC5D therapy (e.g. talquetamab).
* Prior therapy with bispecific antibody therapy within three months
* Prior therapy with gene-modified adoptive cell therapy (e.g. CAR T-cells, NK cells) within three months
* Plasmapheresis within seven days prior to start of study treatment.
* Primary refractory disease.
* Concomitant high dose corticosteroids. Low dose corticosteroids (maximum dose prednisone 10 mg/day or equivalent) are permitted if given for disorders other than myeloma, e.g. adrenal insufficiency, rheumatoid arthritis, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Recommended Dose | Day 1 of treatment through 30 days post last-dose (treatment is until disease progression or withdrawal; estimated to be 1 year from Day 1 of treatment)
  To determine the recommended dose and schedule of mezigdomide and talquetamab in triple class exposed, relapsed and refractory multiple myeloma (RRMM), the dose level where 2 of 6 participants experience a DLT is considered the maximum tolerated dose. The dose level below this will be considered a recommended phase 2 dose. Or if dose level 2 is reached (mezigdomide 1 mg po for 21 out of 28 days) and there are ≤1 DLTs out of 6 participants, then dose level 2 will be considered the recommended phase 2 dose. Data from the secondary outcomes (frequency of adverse events, serious adverse events, and dose-limiting toxicities) will be used for this outcome.

SECONDARY OUTCOMES:
Frequency of adverse events | Day 1 of treatment through 30 days post last-dose (treatment is until disease progression or withdrawal; estimated to be 1 year from Day 1 of treatment)
  Assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, the frequency of AEs will be tabulated by cohort and dose.
Frequency of serious adverse events | Day 1 of treatment through 30 days post last-dose (treatment is until disease progression or withdrawal; estimated to be 1 year from Day 1 of treatment)
  Assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, the frequency of serious AEs will be tabulated by cohort and dose.
Frequency of dose-limiting toxicities (DLT) | Day 1 of treatment through 30 days post last-dose (treatment is until disease progression or withdrawal; estimated to be 1 year from Day 1 of treatment)
  Unacceptable toxicity will be defined as grade 3-4 CRS, grade 3-4 ICANS, and grade 4, treatment-related, non-hematologic adverse events. Assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 when applicable. The frequency and type of DLTs will be tabulated by cohort and dose.
Overall response rate (ORR) | Day 1 of treatment through 2 years post last-dose (estimated total time to be 3 years; treatment is until disease progression or withdrawal)
  Response rate will be according to IMWG criteria. Overall response rate is rate of patients achieving partial response or better.
Progression Free Survival (PFS) | Day 1 of treatment through 2 years post last-dose (estimated total time to be 3 years; treatment is until disease progression or withdrawal)
  Progression-free survival (PFS) is defined as the time from start of treatment to disease progression or death from any cause. Patients who have not progressed or died are censored at the date last known progression-free. Response will be according to IMWG criteria. PFS will be determined from first dose of study drug, according to Kaplan-Meier methodology.
Overall Survival (OS) | Day 1 of treatment through 2 years post last-dose (estimated total time to be 3 years; treatment is until disease progression or withdrawal)
  Overall survival (OS) is defined as the time from start of treatment to death due to any cause or censored at date last known alive. Response will be according to IMWG criteria. OS will be determined from first dose of study drug, according to Kaplan-Meier methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Yee, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Andrew J. Yee, MD, ayee1@mgh.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation